CLINICAL TRIAL: NCT01790620
Title: Impact of a Continuous Dialysis Technique Associated With Adsorption Capacity Membranes in Patients With Sepsis Associated - Acute Kidney Injury.
Brief Title: Impact of CVVHD With Adsorption Capacity Membranes in Septic Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital de Sant Pau (Other)
Responsible Party: Principal Investigator, Joan Sabater Riera, Medical Doctor, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SIRAKI 00-2012; PR 148/12 (Other: Servei de Medicina Intensiva. HUB.)
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Sepsis; Septic Shock; Acute Kidney Injury
Keywords: Sepsis; Septic shock; Acute renal failure; Acute kidney injury; Continuous renal replacement therapies CRRT
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CVVHD-ST150 (Experimental): Patients with sepsis whom present AKI meeting CRRT initiation criteria will be started on CVVHD with PrismafleX eXeed™ II (Hospal) using an ST150SET copolymer of acrylonitrile and sodium methylsulfonate (AN 69) with polyethylenimine treated surface. Anticoagulation of the ST150 set with unfractioned heparin will only be initiated if there´s no clinical contraindication. ST150 set will be changed when clotted and every 24 hours during the first 72 hours of CVVHD. No citrate anticoagulation will be used.
  Interventions: Other: CVVHD
- CVVH-ST150 (Active Comparator): Patients with sepsis whom present AKI meeting CRRT initiation criteria will be started on CVVH with PrismafleX eXeed™ II (Hospal) using an ST150SET copolymer of acrylonitrile and sodium methylsulfonate (AN 69) with polyethylenimine treated surface. Anticoagulation of the ST150 set with unfractioned heparin will only be initiated if there´s no clinical contraindication. ST150 set will be changed when clotted and every 24 hours during the first 72 hours of CVVH. No citrate anticoagulation will be used.
  Interventions: Other: CVVH

INTERVENTIONS:
Other: CVVHD — CVVHD will be used during 72 hours with a prescribed dose of 30 ml/Kg/h Prismasol® 4 as dialysate fluid. Blood flow of 200-250 ml/min, to achieve 12 - 15 L/h will be prescribed. Isovolemic CRRT will be encouraged during this 72 hours if volume overload status is not present. After 72 hours, CVVHD will be continued and dialysate dose (ml/kg/h) will be adjusted to achieve creatinine levels between 80-120 umol/L until patient recovers urine output and / or tolerates intermittent hemodialysis.
  Other Names: Continuous venovenous hemodialysis
  Arms: CVVHD-ST150
Other: CVVH — CVVH will be used during 72 hours with a prescribed dose of 30 ml/Kg/h Prismasol® 4 as reposition fluid. Blood flow of 200-250 ml/min, to achieve 12 - 15 L/h will be prescribed adjusting the adequate percentage of prefilter reinfusion to maintain a theorical filtration fraction between 18-22%. Isovolemic CRRT will be encouraged if volume overload status is not present. After 72 hours, CVVH will be continued and filtration dose (ml/kg/h) will be adjusted to achieve creatinine levels between 80-120 umol/L until patient recovers urine output and / or tolerates intermittent hemodialysis.
  Other Names: Continuous venovenous hemofiltration
  Arms: CVVH-ST150

SUMMARY:
Septic patients with acute kidney injury (SA-AKI) requiring continuous renal replacement therapies (CRRT) present high mortality due to systemic inflammatory response, cytokine liberation, and finally multiorgan dysfunction. Cytokine plasmatic elimination with continuous venovenous hemofiltration (CVVH) presents frequent complications, known as "dialytrauma", and a high resource cost both technical and human. The study primary end-point is to demonstrate a longer filter life with the use of continuous venovenous hemodialysis (CVVHD) respect to CVVH, both modalities employing the same adsorption capacity membrane. As secondary end-points investigators will try to demonstrate less dialytrauma events of CVVHD respect to CVVH. In order to achieve these objectives investigators have designed a proof of concept exploratory trial that will include those patients whom present SA-AKI meeting CRRT initiation criteria. During the first 72 hours investigators will measure plasmatic elimination capacity of main cytokines, and other clinical and prognostic relevant molecules. Investigators will also measure hemodynamic, respiratory, and metabolic parameters. Adverse effects related to CRRT ("dialytrauma") will also be registrated. Finally, investigators will analyze 90 days survival. Demonstration of a minor complication rate (longer filter patency with less dialytrauma events) with a similar immunomodulating capacity and with its consequent lower cost, should settle the based evidence principles that recommend the use of CVVHD asociated to an adsorption capacity membrane in patients with SA-AKI whom need CRRT.

DETAILED DESCRIPTION:
Investigators will warrant a correct protocol application. Study data will be reviewed by an external monitoring committee from the clinical assay research central unit (UCICEC - IDIBELL). Monitors will contrast registered data from the collection data form (CDF) with data from patient´s medical record. All patient´s medical records will be indefinitely saved in electronical format to be reviewed if necessary.

Patients who meet inclusion criteria will be randomized for one of both arms with aleatory assignation using a randomisation sequential (RndSeq) program for Statistical Package for the Social Sciences (SPSS). Adverse events will be reported (in less than 24 hours if severe) to the sponsor center to be properly evaluated. If the severe adverse event (SAE) is finally evaluated by the study board as related to the intervention arm, urgent notification to health authorities must proceed and study should be interrupted until further decision.

As a pilot study of at least 50 cases is advisable in many circumstances (Sim and Lewis, 2012), and we wanted to compare two treatment options, we aimed to recruit at least 100 patients.

Missing data will try to be avoided by an exhaustive patient´s follow up by study investigators. Intention to treat analysis (ITT) will be the main strategy and statistical substitution techniques for missing data will be applied when necessary. Per protocol analysis will also be done to avoid possible bias. Out-of-range results will be identified and processed with adequate statistical techniques.

Data registry has been created to include all variables with written individual data collection forms (DCF). Data will be bedside registered by the study members but final software database registration will be done by the statistics outside investigator who has no contact with patients situation. Cytokines levels will be introduced in DCF when measured (every six months).

Statistical analysis will be done by the statistics investigator who wont have any role in patient´s selection, randomization, or follow up. SPSS v. 18.0 for statistical analysis will be used. Variable distribution will be studied and logarithmic transformation will be used on those variables that don't present normal distribution, presumably cytokine levels. Univariate analysis comparing clinical, demographic, biochemical, metabolic, hemodynamic and respiratory baseline variables between both arms (CVVHD-ST150 and CVVH-ST150), will be done with two-tailed t test for continuous variables and chi-square test for categorical variables. Variables determined several times (T0, T24, T48, T72) will be analysed using a one-way repeated measures ANOVA test in order to demonstrate differences between both arms. Multivariate analysis will be completed to control those clinically relevant confounding variables as well as to discover baseline differences. According to hypothesis and to the dependent variable on study investigators will use a survival analysis (to study mortality) with a cox regression model, or a hierarchic multiple linear regression model when the dependent variable is continuous (for example dialytrauma score). Arm intervention (CVVHD, CVVH) will be considered as the main independent variable adding other control independent variables.

As the study is measuring cytokine levels in five different moments (T0, T24, T48, T72), in order to maximize statistical power and reduce control variables number, the area under the curve (AUC) we´ll be determined for every cytokine and LPS during the first 72 hours. Due to this statistical maneuver investigators will obtain a continuous variable that represents each cytokine level during the biochemical study period (72 hours). To evaluate if the arm intervention improvement in terms of efficacy and safety could be related to cytokine levels during the first 72 hours, a mediation complementary analysis will be done considering cytokine (represented by AUC) as a mediator between the independent variable (intervention arm) and the effect we study.

Data dictionary. ICU: Intensive Care Unit; AKI: Acute Kidney Injury; CRRT: Continuous Renal Replacement Therapies; IL-1β: interleukin 1β; TNF-α: tumor necrosis factor α; IL-6: interleukin 6, IL-10: interleukin 10; IL-4: interleukin 4; CVVH: Continuous Venovenous Hemofiltration; CVVHD: Continuous Venovenous Hemodialysis; SPSS: Statistical Package for the Social Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Less than 72 hours from ICU admission to inclusion
* Clinical diagnosis of Severe Sepsis or Septic shock (SCCM definitions)
* Correct therapeutic initial management of septic process (SSC guidelines)
* Clinical diagnosis of Acute Kidney Injury (ADQI definitions)
* Acute Kidney Injury meeting CRRT initiation criteria (ADQI guidelines)
* Written informed consent from patient or legal surrogates

Exclusion Criteria:

* End Stage Renal Disease(ESRD)
* Received previous CRRT or hemodialysis in the last three months
* Inclusion in other ongoing study
* Coexisting illness with a high probability of death
* Immunosuppression

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Technical CRRT efficiency | 72 hours
  Number of times set was changed.

SECONDARY OUTCOMES:
Safety technical superiority. | 72 hours
  Less adverse events related to CRRT known as "dialytrauma". Red blood cells transfusions related with filter clotting, thrombocytopenia (less than 100.000), hypophosphatemia (less than 0.7 mmol/L), hypokaliemia (less than 3.3 mmol/L), and hypothermia (less than 35.5ºC rectal temperature).
Survival at 90 days after randomization | 90 days.
  Kaplan Meyer survival analysis and cox proportional hazard ratio for death will be both done at 90 days after CRRT initiation.
Immunomodulating capacity | 72 hours
  Cytokine removal: interleukin-1β (IL-1β), tumor necrosis factor α (TNF-α), interleukin 6 (IL-6), interleukin-4 (IL-4), and interleukin-10 (IL-10) levels will be determined in plasma (pre and postfilter) and in ultrafiltrate.
  Determinations will be measured baseline (0hours), and at times 24hours, 48hours, and 72hours. 24h, 48h, and 72h determinations should only be done when ST150 set has been working for at least 6 continuous hours. This means that determinations can be advanced or delayed +/- 4 hours to scheduled time (for example 20 - 28 hours for T24).
Renal depuration capacity. | 72 hours.
  Sieving coefficients for plasma solutes (creatinine, urea, potassium, albumine, magnesium, phosphate, and others) will be determined after measuring blood (pre and postfilter) and ultrafiltrate levels at 24hours, 48 hours, and 72 hours. 24h, 48h, and 72h determinations should only be done when ST150 set has been working for at least 6 continuous hours. This means that determinations can be advanced or delayed +/- 4 hours to scheduled time (for example 20 - 28 hours for T24).
Hemodynamics and respiratory variations. | 72 hours.
  Hemodynamic and respiratory parameters will be registered every hour. Arterial and venous gasometries with arterial lactate will be determined every 6 hours during the first 72 hours.
Clinical efficiency | 90 days
  Days on CRRT. Days on Dialysis. Days of ICU. Days of hospital. Renal recovery at hospital discharge (free from dialysis).

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabater Riera, MD, Principal Investigator — Hospital Universitari de Bellvitge; Xosé L. Pérez Fernández, MD, Study Director — Hospital Universitari de Bellvitge; Antoni Betbesé Roig, MD, Study Director — Hospital de Sant Pau; Jorge Ordoñez Llanos, MD PhD, Study Chair — Hospital de Sant Pau
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

REFERENCES:
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Messer J, Mulcahy B, Fissell WH. Middle-molecule clearance in CRRT: in vitro convection, diffusion and dialyzer area. ASAIO J. 2009 May-Jun;55(3):224-6. doi: 10.1097/MAT.0b013e318194b26c. PMID 19282753
- [Background] Hofmann CL, Fissell WH. Middle-molecule clearance at 20 and 35 ml/kg/h in continuous venovenous hemodiafiltration. Blood Purif. 2010;29(3):259-63. doi: 10.1159/000266483. Epub 2009 Dec 17. PMID 20016150
- [Background] Ricci Z, Ronco C, Bachetoni A, D'amico G, Rossi S, Alessandri E, Rocco M, Pietropaoli P. Solute removal during continuous renal replacement therapy in critically ill patients: convection versus diffusion. Crit Care. 2006;10(2):R67. doi: 10.1186/cc4903. PMID 16646985
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Background] Kellum JA, Johnson JP, Kramer D, Palevsky P, Brady JJ, Pinsky MR. Diffusive vs. convective therapy: effects on mediators of inflammation in patient with severe systemic inflammatory response syndrome. Crit Care Med. 1998 Dec;26(12):1995-2000. doi: 10.1097/00003246-199812000-00027. PMID 9875910
- [Background] Saudan P, Niederberger M, De Seigneux S, Romand J, Pugin J, Perneger T, Martin PY. Adding a dialysis dose to continuous hemofiltration increases survival in patients with acute renal failure. Kidney Int. 2006 Oct;70(7):1312-7. doi: 10.1038/sj.ki.5001705. Epub 2006 Jul 19. PMID 16850022
- [Background] RENAL Replacement Therapy Study Investigators; Bellomo R, Cass A, Cole L, Finfer S, Gallagher M, Lo S, McArthur C, McGuinness S, Myburgh J, Norton R, Scheinkestel C, Su S. Intensity of continuous renal-replacement therapy in critically ill patients. N Engl J Med. 2009 Oct 22;361(17):1627-38. doi: 10.1056/NEJMoa0902413. PMID 19846848
- [Background] VA/NIH Acute Renal Failure Trial Network; Palevsky PM, Zhang JH, O'Connor TZ, Chertow GM, Crowley ST, Choudhury D, Finkel K, Kellum JA, Paganini E, Schein RM, Smith MW, Swanson KM, Thompson BT, Vijayan A, Watnick S, Star RA, Peduzzi P. Intensity of renal support in critically ill patients with acute kidney injury. N Engl J Med. 2008 Jul 3;359(1):7-20. doi: 10.1056/NEJMoa0802639. Epub 2008 May 20. PMID 18492867
- [Background] Maynar Moliner J, Honore PM, Sanchez-Izquierdo Riera JA, Herrera Gutierrez M, Spapen HD. Handling continuous renal replacement therapy-related adverse effects in intensive care unit patients: the dialytrauma concept. Blood Purif. 2012;34(2):177-85. doi: 10.1159/000342064. Epub 2012 Oct 24. PMID 23095418
- [Background] Ronco C, Bellomo R, Homel P, Brendolan A, Dan M, Piccinni P, La Greca G. Effects of different doses in continuous veno-venous haemofiltration on outcomes of acute renal failure: a prospective randomised trial. Lancet. 2000 Jul 1;356(9223):26-30. doi: 10.1016/S0140-6736(00)02430-2. PMID 10892761
- [Background] Rogiers P, Zhang H, Smail N, Pauwels D, Vincent JL. Continuous venovenous hemofiltration improves cardiac performance by mechanisms other than tumor necrosis factor-alpha attenuation during endotoxic shock. Crit Care Med. 1999 Sep;27(9):1848-55. doi: 10.1097/00003246-199909000-00024. PMID 10507609
- [Background] De Vriese AS, Colardyn FA, Philippe JJ, Vanholder RC, De Sutter JH, Lameire NH. Cytokine removal during continuous hemofiltration in septic patients. J Am Soc Nephrol. 1999 Apr;10(4):846-53. doi: 10.1681/ASN.V104846. PMID 10203370
- [Background] Bozza FA, Salluh JI, Japiassu AM, Soares M, Assis EF, Gomes RN, Bozza MT, Castro-Faria-Neto HC, Bozza PT. Cytokine profiles as markers of disease severity in sepsis: a multiplex analysis. Crit Care. 2007;11(2):R49. doi: 10.1186/cc5783. PMID 17448250
- [Background] Gogos CA, Drosou E, Bassaris HP, Skoutelis A. Pro- versus anti-inflammatory cytokine profile in patients with severe sepsis: a marker for prognosis and future therapeutic options. J Infect Dis. 2000 Jan;181(1):176-80. doi: 10.1086/315214. PMID 10608764
- [Background] Marshall JC, Foster D, Vincent JL, Cook DJ, Cohen J, Dellinger RP, Opal S, Abraham E, Brett SJ, Smith T, Mehta S, Derzko A, Romaschin A; MEDIC study. Diagnostic and prognostic implications of endotoxemia in critical illness: results of the MEDIC study. J Infect Dis. 2004 Aug 1;190(3):527-34. doi: 10.1086/422254. Epub 2004 Jul 2. PMID 15243928
- [Background] Gibney N, Hoste E, Burdmann EA, Bunchman T, Kher V, Viswanathan R, Mehta RL, Ronco C. Timing of initiation and discontinuation of renal replacement therapy in AKI: unanswered key questions. Clin J Am Soc Nephrol. 2008 May;3(3):876-80. doi: 10.2215/CJN.04871107. Epub 2008 Mar 5. PMID 18322044
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356